CLINICAL TRIAL: NCT03431753
Title: Early and Accurate Detection of Prostate Cancer in General Practice Using Novel Molecular Biomarkers and Multiparametric MR Imaging.
Brief Title: Early and Accurate Detection of Prostate Cancer in General Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Aarhus University Hospital (Other)
Collaborators: Regional Hospital Holstebro (Other); University of Aarhus (Other); Central Denmark Region (Other); Karolinska Institutet (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRIMA
Record Dates: First submitted 2017-12-21; First posted 2018-02-13 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer; Prostate Neoplasm; Prostate Adenocarcinoma
Keywords: STHLM3-test; prostate cancer; MR-imaging; MR-targeted biopsy; MRI; Novel biomarkers; Genetic screening
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSA, STHLM3 and mpMRI for PC detection (Experimental): mpMRI, and if suspect MR-targeted prostate biopsy, in men with increased PC risk as judged from the STHLM3 test and/or an elevated prostate specific antigen test.
  Interventions: Diagnostic Test: PSA, STHLM3 and mpMRI for PC detection

INTERVENTIONS:
Diagnostic Test: PSA, STHLM3 and mpMRI for PC detection — Men who request a prostate specific antigen test from their general practitioner will be offered study participation.
  Men with increased PC risk as judged from the STHLM3 test and/or an elevated PSA test will be offered an mpMRI examination.

SUMMARY:
Prostate cancer (PC) is the most common malignancy (4500 new cases/year) and the second leading cause of cancer-associated mortality (1200 deaths/year) among men in Denmark. PC is generally diagnosed on the basis of an elevated prostate specific antigen blood test followed by transrectal ultrasound (TRUS)-guided prostate biopsy.

This study aims to test early detection of PC in general practice, using the STHLM3 model with superior specificity and sensitivity for clinically significant PC, combined with multiparametric magnetic resonance imaging (mpMRI) of the prostate and MR guided biopsy.

DETAILED DESCRIPTION:
While early stage PC can be cured by surgery or radiation therapy, advanced PC is incurable and associated with high morbidity and mortality. Early detection is critical to save lives, but many newly diagnosed PCs are in reality non-aggressive and will not affect the patient's life or health, even if left untreated. There is an urgent need to replace current clinical practice with a more accurate diagnostic approach that can ensure early detection of aggressive PC while curable, reduce unnecessary prostate biopsies incl. risk of sepsis and reduce overdiagnosis/-treatment of indolent PC.

New molecular biomarkers applied in general practice, serving as a pre-selection test for follow-up, and accurate and patient-friendly MR-imaging and MR-targeted biopsy at the hospital may help to solve these problems.

In this study the investigators will assess the clinical utility of combining genetic risk testing and plasma protein markers (STHLM3 test) in general practice with mpMRI and MR-guided in bore biopsy (MRGB) for early PC detection in a biopsy naïve population.

ELIGIBILITY:
Inclusion Criteria:

* aged 50-69 years
* no previous pelvic cancer
* no previous prostate biopsy
* no previous elevated PSA results
* informed consent from the participant

Exclusion Criteria:

* palpable prostatae tumor by digital rectal examination
* previously diagnosed with/or treated for an urogenital cancer disease
* contraindications to 3 T MRI
* known severe renal impairment with estimated glomerular filtration rate <30 ml / min

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of PC suspicious lesions detected by mpMRI based on the STHLM3 test vs. the prostate specific antigen test. | 24 months
  Evaluation of the proportion of patients identified with PC suspicious lesions at mpMRI based on the STHLM3 vs. the prostate specific antigen test.

SECONDARY OUTCOMES:
Proportion of PC diagnoses detected in the study population based on the STHLM3 test vs. the prostate specific antigen test. | 24 months
  Evaluation of the proportion of total PCs and clinically significant PCs diagnosed with MR guided biopsy as a function of the primary tests.
Compare results from clinical study with current clinical practice. | 24 months
  Comparison of the results from the clinical study with the number of prostate specific antigen tests, TRUS-biopsies, indolent and significant PCs detected by current clinical practice, using health register data from general practices not taking part in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Bodil G. Pedersen, MD, PhD, Principal Investigator — Department of Radiology, Aarhus University Hospital; Karina D. Sørensen, Professor, Principal Investigator — Dept. of Molecular Medicine (MOMA) at Aarhus University Hospital
Locations (1):
- General Practice, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No